CLINICAL TRIAL: NCT03912948
Title: Prospective Cohort Study Assessing Chronic Pain in Patients With Thoracic Blocks Following Minor Surgery for Breast Cancer.
Brief Title: Chronic Pain and Minor Breast Cancer Surgery
Acronym: DCPO Sein
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: CNIL-2033408
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-04

CONDITIONS: Surgery; Breast Cancer; Pain, Postoperative; Pain, Chronic
Keywords: regional analgesia techniques; breast cancer surgery; conservative surgery
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most frequent in women. Early diagnosis and recent treatments have improved overall mortality. However, chronic pain (pain lasting more than 3 months after surgery) remains a public health problem with impact on quality of life for these patients. The incidence of pain has been reported up to 25 to 60% of patients in the literature, even many years after a radical mastectomy. The neuropathic component of the pain is usually underestimated. In a prospective cohort study we have demonstrated that 43% of patient needed on average 5mg of morphine intravenously in the recovery room after a conservative breast cancer surgery, despite a multimodal regimen of analgesic drugs. In the same study, 40% of patients reported persistent pain 3 months after the surgery. To improve the analgesia in such a population, we decided to introduce regional analgesia technique (serratus block) systematically. This became our gold standard in our daily practice. We would like to assess the efficacy of such regional analgesia techniques on opioids consumption in the recovery room and the incidence of pain 3 months after conservative breast cancer surgery.

DETAILED DESCRIPTION:
This is a prospective observational study assessing the interest of preoperative thoracic block (injection of local anesthetic around the serratus muscle under ultrasound guidance) in the prevalence of chronic pain 3 months after a conservative breast cancer surgery.

Information on the present survey was given during pre-operative consultation and signed informed consent was obtained to enter the study.

The management of patients undergoing minor surgery for breast cancer is standardized within our department and reported in our previous study. After starting the induction of anesthesia and insertion of a laryngeal mask, a regional analgesia technique was performed under ultrasonography. Twenty ml of ropivacaine 3.75mg/ml were injected under the serratus muscle, at the lateral edge of the minor pectoralis muscle. In the absence of contraindications, multimodal analgesia consisted of paracetamol, non-steroidal anti-inflammatory drugs and nefopam. Postoperative intravenous morphine titration was possible in patients presenting a pain score >3/10 (numeric pain intensity scale from 0 = no pain to 10 = maximum imaginable pain) in the recovery room. If 0.1mg/kg of morphine did not permit to alleviate pain, ketamine titration was initiated by the anesthesiologist.

The incidence of patients that required opioids titration in the recovery room (and the dose injected) was recorded.

The questionnaire sent to the patients 3 months after their surgery was mainly composed of closed questions. This questionnaire included pain score, location of pain, analgesic drugs consumption, neuropathic component (self-administered questionnaire derived from the Neuropathic Pain 4 Questions - DN4 questionnaire), impact of quality of life using the Brief Pain Inventory.

ELIGIBILITY:
Inclusion Criteria:

* women
* > 18 years old
* with "American Society of Anesthesiologists-ASA" physical status 1 to 3
* with unilateral breast cancer adenocarcinoma treated surgically by conservative tumorectomy associated or not to sentinel lymph node dissection on an ambulatory basis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women >18yrs old, with ASA physical status 1 to 3, with unilateral breast adenocarcinoma treated surgically by conservative tumorectomy ± associated to sentinel lymph node dissection on an ambulatory basis.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of chronic pain | 3 months
  To assess the number (%) of patients presenting persistent pain 3 months after minor breast cancer surgery

SECONDARY OUTCOMES:
Incidence of pain | 3 months
  incidence of pain and mean dose of morphine injected in the recovery room, percentage of neuropathic component among patients presenting persistent pain at 3 months; impact of pain on quality of life, risk factors to develop postoperative persistent pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius Regaud - IUCT-Oncopole, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No
Will not be shared

REFERENCES:
- [Result] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Result] Fuzier R, Puel F, Izard P, Sommet A, Pierre S. Prospective cohort study assessing chronic pain in patients following minor surgery for breast cancer. J Anesth. 2017 Apr;31(2):246-254. doi: 10.1007/s00540-016-2288-9. Epub 2016 Nov 24. PMID 27885426
- Available data/document: Web site for patient information on studies bases on patients data (RGPD) — https://www.iuct-oncopole.fr/recherches-necessitant-une-reutilisation-de-donnees